CLINICAL TRIAL: NCT00008060
Title: Fluorouracil, Oxaliplatin and Irinotecan: Use and Sequencing: A Randomized Trial to Assess the Role of Irinotecan and Oxaliplatin in Advanced Colorectal Cancer
Brief Title: Combination Chemotherapy in Treating Patients With Unresectable Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068372; MRC-CR08-FOCUS; EU-20038; ISRCTN79877428
Record Dates: First submitted 2001-01-06; First posted 2003-01-27 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2002-03

CONDITIONS: Colorectal Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Neoplasms; Rectal Neoplasms | interventions — Folfox protocol; Fluorouracil; Irinotecan; Leucovorin; Oxaliplatin

INTERVENTIONS:
Drug: FOLFIRI regimen
Drug: FOLFOX regimen
Drug: fluorouracil
Drug: irinotecan hydrochloride
Drug: leucovorin calcium
Drug: oxaliplatin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which regimen of combination chemotherapy is more effective for advanced colorectal cancer.

PURPOSE: Randomized phase III trial to compare the effectiveness of fluorouracil combined with leucovorin and either irinotecan or oxaliplatin in treating patients who have unresectable metastatic colorectal cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of combination chemotherapy comprising fluorouracil (5-FU) with leucovorin calcium (CF) and either irinotecan (CPT-11) or oxaliplatin vs standard sequential single-agent therapy comprising 5-FU with CF followed by CPT-11 in patients with unresectable metastatic colorectal cancer.
* Determine whether combination chemotherapy is best used as first-line therapy or reserved for second-line therapy after progression on first-line single-agent therapy in these patients.
* Compare the efficacy and toxicity of an irinotecan-containing regimen vs an oxaliplatin-containing regimen in these patients.
* Compare the overall survival, progression-free survival, and quality of life of patients treated with these regimens.
* Compare the safety and toxicity of these regimens in these patients.

OUTLINE: This is a randomized, open-label, multicenter study. Patients are randomized to one of five treatment arms.

* Arm I (standard therapy): Patients receive first-line chemotherapy comprising leucovorin calcium IV over 2 hours on day 1 followed by fluorouracil IV continuously over 46 hours on days 1-2 every 14 days. Patients with progressive disease then receive second-line therapy comprising irinotecan IV over 90 minutes on day 1 every 21 days.
* Arm II: Patients receive first-line chemotherapy as in arm I. Patients with progressive disease then receive second-line therapy comprising irinotecan IV over 30 minutes and leucovorin calcium IV over 2 hours on day 1 and fluorouracil IV continuously over 46 hours on days 1-2 every 14 days.
* Arm III: Patients receive first-line chemotherapy comprising irinotecan, leucovorin calcium, and fluorouracil as in second-line therapy of arm II.
* Arm IV: Patients receive first-line chemotherapy as in arm I. Patients with progressive disease then receive second-line therapy comprising leucovorin calcium IV and oxaliplatin IV over 2 hours on day 1 followed by fluorouracil IV continuously over 46 hours on days 1-2 every 14 days.
* Arm V: Patients receive first-line chemotherapy comprising leucovorin calcium, oxaliplatin, and fluorouracil as in second-line therapy of arm IV.

Treatment continues in all arms in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline, at weeks 6 and 12, and then every 12 weeks thereafter.

PROJECTED ACCRUAL: A total of 2,100 patients (700 in arm I and 350 each in arms II-V) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed metastatic adenocarcinoma of the colon or rectum

  * Unresectable disease
* Measurable or evaluable disease
* No partial or complete bowel obstruction

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* WHO 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 4,000/mm^3
* Platelet count greater than 150,000/mm^3

Hepatic:

* Bilirubin less than 1.25 times upper limit of normal (ULN)
* Alkaline phosphatase less than 5 times ULN
* AST or ALT less than 3 times ULN
* No Gilbert's syndrome or other congenital abnormality of biliary transport (e.g., Crigler-Najjar syndrome or Dubin-Johnson syndrome)

Renal:

* Creatinine clearance greater than 50 mL/min OR
* Glomerular filtration rate normal

Other:

* Not pregnant
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other uncontrolled medical illness
* No other prior or concurrent malignancy that would preclude study entry
* No chronic diarrhea or inflammatory bowel disease
* No grade 2 or greater pre-existing neuropathy

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* At least 6 months since prior adjuvant chemotherapy
* Prior adjuvant fluorouracil allowed
* No prior chemotherapy for metastatic disease
* No prior oxaliplatin or irinotecan

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* No prior transplantation surgery requiring immunosuppressive therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-05; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew T. Seymour, MA, MD, FRCP, Study Chair — Medical Research Council
Locations (1):
- Medical Research Council Clinical Trials Unit, London, England, United Kingdom

REFERENCES:
- [Background] Richman SD, Chambers P, Seymour MT, Daly C, Grant S, Hemmings G, Quirke P. Intra-tumoral heterogeneity of KRAS and BRAF mutation status in patients with advanced colorectal cancer (aCRC) and cost-effectiveness of multiple sample testing. Anal Cell Pathol (Amst). 2011;34(1-2):61-6. doi: 10.3233/ACP-2011-0005. PMID 21483104
- [Result] Braun MS, Richman SD, Thompson L, Daly CL, Meade AM, Adlard JW, Allan JM, Parmar MK, Quirke P, Seymour MT. Association of molecular markers with toxicity outcomes in a randomized trial of chemotherapy for advanced colorectal cancer: the FOCUS trial. J Clin Oncol. 2009 Nov 20;27(33):5519-28. doi: 10.1200/JCO.2008.21.6283. Epub 2009 Oct 26. PMID 19858398
- [Result] Richman SD, Seymour MT, Chambers P, Elliott F, Daly CL, Meade AM, Taylor G, Barrett JH, Quirke P. KRAS and BRAF mutations in advanced colorectal cancer are associated with poor prognosis but do not preclude benefit from oxaliplatin or irinotecan: results from the MRC FOCUS trial. J Clin Oncol. 2009 Dec 10;27(35):5931-7. doi: 10.1200/JCO.2009.22.4295. Epub 2009 Nov 2. PMID 19884549
- [Result] Seymour MT, Maughan TS, Ledermann JA, Topham C, James R, Gwyther SJ, Smith DB, Shepherd S, Maraveyas A, Ferry DR, Meade AM, Thompson L, Griffiths GO, Parmar MK, Stephens RJ; FOCUS Trial Investigators; National Cancer Research Institute Colorectal Clinical Studies Group. Different strategies of sequential and combination chemotherapy for patients with poor prognosis advanced colorectal cancer (MRC FOCUS): a randomised controlled trial. Lancet. 2007 Jul 14;370(9582):143-152. doi: 10.1016/S0140-6736(07)61087-3. PMID 17630037
- [Result] Maughan T: Fluorouracil (FU), oxaliplatin (OX), CPT-11 (irinotecan, Ir), use and sequencing, in advanced colorectal cancer (ACRC): the UK MRC FOCUS (CR08) trial. [Abstract] American Society of Clinical Oncology 2005 Gastrointestinal Cancers Symposium, 27-29 January 2005, Miami, Florida. A-165, 2005.
- [Result] Seymour MT: Fluorouracil, oxaliplatin and CPT-11 (irinotecan), use and sequencing (MRC FOCUS): a 2135-patient randomized trial in advanced colorectal cancer (ACRC). [Abstract] J Clin Oncol 23 (Suppl 16): A-3518, 250s, 2005.
- [Result] Seymour M: An update on the MRC FOCUS/CR08 trial: the first 300 patients. [Abstract] Br J Cancer 85 (suppl 1): A-P45, 44, 2001.